CLINICAL TRIAL: NCT00296582
Title: Simultaneous Gastric Motor Function Measurement in Dyspepsia And Normal Subjects Ingesting a Solid-Liquid Meal
Brief Title: Gastric Motor Function Measurement in Dyspepsia and Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Hack Jae Kim, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 65-06
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Gastric Motor Function Measurement

SUMMARY:
This study is being done to measure the functions of the stomach after eating a meal and to develop a new method that will simultaneously measure both gastric emptying and the relaxation of the stomach after a meal using nuclear medicine testing. This would make the testing more convenient for patients and will also offer better understanding of these two gastric functions.

ELIGIBILITY:
Inclusion criteria:

Dyspeptic Subjects:

* Recurrent episodes of upper abdominal pain or discomfort including early satiety, fullness, bloating, or nausea for at least 3 months in the prior year.
* A baseline impaired satiety test (maximum tolerated volume 25% of normal or 1000cc).
* No evidence on esophagogastroduodenoscopy of erosions, peptic ulcer, pyloric obstruction, esophagitis or malignancy in the prior 3 years.

All Subjects:

* No history suggestive of small bowel obstruction.

Exclusion criteria

* No structural or metabolic diseases/conditions that affect the gastrointestinal system.
* Unable to stop medications 48 hours prior to the study that:

  * Alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, SSRI and newer antidepressants.
  * Analgesic drugs including opiates, NSAID, COX 2 inhibitors
  * Systemic antifungal drugs
  * Carbamazepine, glucocorticoids, phenobarbital, phenytoin, rifampin, but also grapefruit juice.
  * Benzodiazepines NOTE: Low stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection and birth control pills or depot injections are permissible.
* Female subjects who are pregnant or breast feeding.
* Significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study.
* Subjects who have participated in another clinical study within the past 30 days.
* Previous gastric or intestinal surgery (except appendectomy , cholecystectomy or hysterectomy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial gastric volumes (Gastric accommodation)

SECONDARY OUTCOMES:
T1/2 of gastric emptying of solid
Maximum tolerated volume
Individual postprandial symptom scores

CONTACTS AND LOCATIONS:
Overall Officials: H. Jae Kim, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States